CLINICAL TRIAL: NCT04710056
Title: Expanded Access to REGN4461 for Patients With Lipodystrophy or Monogenic Obesity With Complications of Leptin Deficiency or Deficient Leptin Signaling
Status: Available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R4461-LEPR
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Lipodystrophy
Keywords: Leptin (LEP); Leptin Receptors (LEPR)
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: REGN4461
  Other Names: mibavademab

SUMMARY:
Provide Expanded Access to REGN4461 for patients with lipodystrophy or monogenic obesity with complications of leptin deficiency or deficient leptin signaling

DETAILED DESCRIPTION:
Expanded Access requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications. Availability will depend on location.

Age Groups: Child, Adult, Older Adult